CLINICAL TRIAL: NCT02618876
Title: Nalbuphine as an Adjuvant to Caudal Bupivacaine for Postoperative Analgesia in Children Undergoing Hypospadias Repair
Brief Title: Effect of Caudal Nalbuphine on Postoperative Analgesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Bakri, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB 000087145
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nalbuphine group (Active Comparator): 30 children will be given Caudal Bupivacaine plus Nalbuphine.
  Interventions: Drug: Nalbuphine plus Bupivacaine
- Control group (Other): 30 children will be given Caudal Bupivacaine.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Nalbuphine plus Bupivacaine — Addition of caudal Nalbuphine to the standard Bupivacaine
  Arms: Nalbuphine group
Drug: Bupivacaine — Caudal Bupivacaine is the standard of care will be considered as a control
  Arms: Control group

SUMMARY:
Nalbuphine as an adjuvant to bupivacaine caudal anesthesia for postoperative analgesia in children undergoing Hypospadias repair.

2 groups, 30 patients each

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing elective Hypospadias repair
* with American Society of Anesthesiologists (ASA) physical status I
* age 2-10 years

Exclusion Criteria:

* Coagulation disorder
* allergy to study medications
* major malformations of the lower spine or meninges or any cutaneous or subcutaneous lesion at the site of injection.

Ages: 2 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity Measured by Face, Legs, Activity, Cry & consolability (FLACC) pain scale | During 24 h in the postoperative period

SECONDARY OUTCOMES:
Cortisol level | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt